CLINICAL TRIAL: NCT02667132
Title: Granulomatous Mastitis Current Approach and Treatment (Multicentric Study) Granulomatous Mastitis Working Group
Brief Title: Granulomatous Mastitis Current Approach and Treatment
Status: Completed | Type: Observational
Sponsor: Granulomatous Mastitis Working Group (Other)
Responsible Party: Sponsor
Other Study IDs: GranulomatousMWG
Record Dates: First submitted 2016-01-11; First posted 2016-01-28 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Granulomatous, Mastitis
Keywords: Granulomatous, Mastitis; C17.800.090.968.400; C13.703.844.603.400
MeSH Terms: conditions — Granulomatous Mastitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- medical treatment: In this study, patient's data will be retrospectively obtained by recording the data in patients' files and electronic records. The data includes the determined parameters by the study group of GM and the data will be recorded in an excel file that includes specific columns of the following entries: patients' age, diagnosis, secondary disease, diagnosis methods, treatments, recurrence, the risk factors that may cause the disease (smoking, using oral contraceptive, breast infection etc.). antibiotic, immunosuppressive drugs, methotrexate
- surgical treatment: lumpectomy, mastectomy, abscess drainage
- surgical+medical treatment: first medical, after surgical treatment or first surgical, after medical treatment

SUMMARY:
The aim of this study was to retrospectively review the granulomatous mastitis and evaluated current approach and treatment.

HYPOTHESIS Although there is no common protocol for the treatment and management process of GM, the ternary treatment (medical treatment following by surgical procedure, Steroid+Antibiotic and surgical procedure, respectively) is considered as the most successful treatment approach.

DETAILED DESCRIPTION:
INTRODUCTION Granulomatous mastitis (GM) is a rare inflammatory disease of the breast which generally affects young parous women. It was emphasized that lactation and using oral contraceptive are considered among the predisposing factors of the disease. GM is firstly identified in 1972, and it is considered as an important disease because it is a great mimicker of breast carcinoma.

The form of treatments involves corticosteroids, antibiotics and general surgical resections including mastectomy. Furthermore, a preferred form of treatment has not been defined yet. Also, there are not enough data showing the results of using antibiotics. Since GM is a rare disease, there is no common consensus for the diagnosis and treatment of GM. The uncertainties about the distinct diagnosis, determining the form and term of treatment, the order of treatment if necessary, as well as what medical specialties need to involve in the treatment process still remain. Therefore, all these uncertainties cause a difficulty to manage the treatment process by physicians. Furthermore, since there is no enough study on GM and only limited case reports was presented in the literature, the success of treatment process is associated with the experience of treatment center. Therefore, there is a clear need for multicentric study that compares different approaches of the treatment process with the enough number of cases.

DATA COLLECTION In this study, patient's data will be retrospectively obtained by recording the data in patients' files and electronic records. The data includes the determined parameters by the study group of GM and the data will be recorded in an excel file that includes specific columns of the following entries: patients' age, diagnosis, secondary disease, diagnosis methods, treatments, recurrence, the risk factors that may cause the disease (smoking, using oral contraceptive, breast infection etc.). A shared excel file at the following website http://sanko.edu.tr/GranulamatozMastit has been created to record the data simultaneously. Each researcher can add the data at the file by using username and password. After data collection, the data will be presented mean+StDv. Statistical analysis will include Mann-Whitney U test, student's t test and chi-square test and statistical significance will set at P< 0.05. The treatment group in this study will be divided as medical, surgical and medical+surgical and the comparison among these groups will be conducted to reach the aims determined in expected outcomes section. The sample size and power analysis were conducted and the results indicated that at least 100 samples in each group are required to achieve the statistical significance at P< 0.05 with 90% power. The estimated total cases are expected over 400 cases.

EXPECTED OUTCOMES

1. Potential etiologies will be investigated.
2. The results will shed light on the optimal management method for patients with GM.
3. The treatment duration and order will be revealed.
4. Treatment and management algorithm will be created.
5. The hypothesis on the success of ternary treatment approach will be tested.
6. Creation of a prognostic index for GM will be tried.
7. Since a multicentric study is planned, experiences and results from different centers will be investigated.
8. Since the study will be multicentric with enough number of cases, the true statistical results will be obtained.
9. Among which medical specialties should be involved in communication during the determination of diagnosis and treatment will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* All Granulomatous Mastitis

Exclusion Criteria:

* Breast Carcinoma

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: from 18 to 90 years womens with Granulomatous Mastitis
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Granulomatous Mastitis Working Group | dec 2015 start data collection, February 2016 The primary outcome statement - April 2016 end up study
  The data includes the determined parameters by the study group of GM and the data will be recorded in an excel file that includes specific columns of the following entries: patients' age, diagnosis, secondary disease, diagnosis methods, treatments, recurrence, the risk factors that may cause the disease. A shared excel file at the following website http://sanko.edu.tr/GranulamatozMastit has been created to record the data simultaneously. Each researcher can add the data at the file by using username and password. After data collection, statistical analysis will include Mann-Whitney U test, student's t test and chi-square test and statistical significance will set at P< 0.05.The sample size and power analysis were conducted and the results indicated that at least 100 samples in each group are required to achieve the statistical significance at P< 0.05 with 90% power. The estimated total cases are expected over 400 cases.

CONTACTS AND LOCATIONS:
Overall Officials: Atilla Soran, Professor, Study Director — Granulomatous Mastitis Working Group
Locations (1):
- Atilla Soran, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
DATA COLLECTION A shared excel file at the following website http://sanko.edu.tr/GranulamatozMastit has been created to record the data simultaneously. Each researcher can add the data at the file by using username and password. After data collection, the data will be presented mean+StDv. Statistical analysis will include Mann-Whitney U test, student's t test and chi-square test and statistical significance will set at P< 0.05. The treatment group in this study will be divided as medical, surgical and medical+surgical and the comparison among these groups will be conducted to reach the aims determined in expected outcomes section. The sample size and power analysis were conducted and the results indicated that at least 100 samples in each group are required to achieve the statistical significance at P< 0.05 with 90% power. The estimated total cases are expected over 400 cases.

REFERENCES:
- [Result] Lee JH, Oh KK, Kim EK, Kwack KS, Jung WH, Lee HK. Radiologic and clinical features of idiopathic granulomatous lobular mastitis mimicking advanced breast cancer. Yonsei Med J. 2006 Feb 28;47(1):78-84. doi: 10.3349/ymj.2006.47.1.78. PMID 16502488
- [Result] Kok KY, Telisinghe PU. Granulomatous mastitis: presentation, treatment and outcome in 43 patients. Surgeon. 2010 Aug;8(4):197-201. doi: 10.1016/j.surge.2010.02.002. Epub 2010 Mar 6. PMID 20569938